CLINICAL TRIAL: NCT01294943
Title: Evaluating the Effectiveness of the Tongue Cleaner in Patients Wholly or Partially Dependent Care
Brief Title: Evaluating the Effectiveness of the Tongue Cleaner in Critical Patients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Paulo Sergio da Silva Santos, DDS, MD, PhD, University of Sao Paulo
Other Study IDs: Bauru School of Dentistry, USP
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Oral Infection; Ventilator-associated Pneumonia
Keywords: Intensive Care Units; Biofilms; Tongue; Infection; Pneumonia/Aspiration
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tongue biofilm
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tongue cleaner: Use of the tongue cleaner (TePe ®) to remove the tongue biofilm in patients on mechanical ventilation.
  Interventions: Device: Tongue cleaner

INTERVENTIONS:
Device: Tongue cleaner — Use of the tongue cleaner (TePe ®) to remove the tongue biofilm in patients on mechanical ventilation.

SUMMARY:
The concern with oral infection and its systemic repercussions is old, many studies have been undertaken to establish this relationship more precisely. One of the areas mouth still little studied in this regard is the colonization of language within this universe of the oral microbiota colonization and how this may affect the general state of health care-dependent individuals.

This research aims to evaluate the efficiency of a tongue cleaning device and its potential impacts on infectious patients fully or partially dependent care hospital.

Patients admitted to intensive care units and inpatient units will be evaluated, divided into two groups: Study Group (SG) - Patients who receive oral hygiene using the tongue cleaning device, and Control Group (CG) - Patients who are cared for according to the routine of hospital nursing.

DETAILED DESCRIPTION:
Patients admitted to intensive care units and inpatient units will be evaluated, divided into two groups: Study Group (SG) - Patients who receive oral hygiene using the tongue cleaning device, and Control Group (CG) - Patients who are cared for According to the routine of hospital nursing.

The criteria for inclusion of elements of the research will follow the criteria of dependence of patients on mechanical ventilation, if they are or not. Patients fully or partially dependent care are patients who can not make your oral hygiene alone and dependent on another individual to do so, if a hospital staff member health. Exclusion criteria will be based on condition of dependency of the patient, intubation period under 48 hours and if one refuses to participate in the research.

Patients will first be evaluated by a dentist, doctor and nursing, which together decide on the inclusion of patients in the study based on the criterion of seriousness of the patient by APACHE. The assessment will follow the clinical criterion of presence or absence of tongue biofilm (Adachi 2005), and the collection swab with biofilm lingual to perform culture and sensitivity. These assessments take place twice within five days, being held in the first and fifth days. During this period the patients participating in the GE will hygienic tongue using tongue cleaner (Tepe ®) and other standardized oral hygiene care by the nursing team previously coached by dentist. CG patients receive the standard oral hygiene care with a spatula and gauze soaked in mouthwash and tongue will not use the tongue cleaner.

For the assessment of plaque and tongue of sample qualitative material for culture and sensitivity attend three calibrated dentists.

For this study 25 patients will be assessed for EG and 25 for GC, a total of 50 patients evaluated, and 100 samples of material collected.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion of elements of the research will follow the criteria of dependence of patients on mechanical ventilation they are or not. Patients fully or partially dependent care are patients who can not make your oral hygiene alone and dependent on another individual to do so, if a hospital staff member health.

Exclusion Criteria:

* Condition of not being dependent on the patient
* Intubation period under 48 hours
* If one refuses to participate in the research

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing intubation in the intensive care unit
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Cruz, São Paulo, São Paulo, Brazil